CLINICAL TRIAL: NCT02429778
Title: Reducing Late-Life Anxiety and Improving Functioning With Self-Directed Relaxation
Brief Title: Relaxation Treatment for Anxiety in Adults Aged 60 or Older
Acronym: BREATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Christine Gould, Instructor (affiliated), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOU0001APR; 22277 (Other Grant/Funding Number: Brain and Behavior Research Foundation)
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Behavioral Intervention (relaxation, breathing, activity engagement)
Oversight: Data Monitoring Committee: No

ARMS (2):
- BREATHE (Experimental): 4 weeks DVD-delivered relaxation intervention program called breathe. The experimental intervention includes progressive muscle relaxation, diaphragmatic breathing, and home practice of the skills. Following the 4 weeks of treatment, participants will be asked to continue to practice at home for 4 weeks.
  Interventions: Behavioral: Diaphragmatic Breathing; Behavioral: Progressive Muscle Relaxation
- Wait List (No Intervention): 8 week wait list period. Participants assigned to wait list will have the opportunity to receive BREATHE arm after 8 weeks if interested.

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing — Deep or diaphragmatic breathing is taught prior to relaxation.
  Other Names: Deep breathing
  Arms: BREATHE
Behavioral: Progressive Muscle Relaxation — Tensing and releasing muscle groups in a specified order to help reduce tension and anxiety.
  Other Names: Progressive Relaxation Training
  Arms: BREATHE

SUMMARY:
The PI developed a self-directed program to treat late-life anxiety called Breathing, Relaxation, and Education for Anxiety Treatment in the Home Environment (BREATHE). This program consists of weekly video lessons that participants watch on digital video disc (DVD) along with weekly telephone check-ins. In BREATHE participants will learn two behavioral interventions: diaphragmatic breathing and progressive muscle relaxation (PMR). The purpose of the study is to examine whether the self-directed BREATHE program is superior to a wait list control in reducing anxiety in older adults with anxiety disorders. For those assigned to wait list control, they will be offered opportunity to participate in BREATHE treatment after 8 weeks of wait list.

ELIGIBILITY:
Inclusion Criteria:

* Participants have a diagnosis of an anxiety disorder, specifically, Generalized Anxiety Disorder, Panic Disorder, Agoraphobia, Social Anxiety Disorder or Anxiety Disorder Unspecified/Other Specified).
* Participants speak English.

Exclusion Criteria:

* Diagnosis of Dementia
* Probable presence of significant cognitive impairment according to a brief cognitive screen
* Serious mental illness (schizophrenia, psychosis, bipolar disorder)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Gould, PhD, Principal Investigator — VA Palo Alto/Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deideintified data will be shared upon reasonable request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BREATHE | Wait List
Started | 20 | 20
Completed | 13 | 20
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BREATHE | Wait List | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.40 (6.77) | 69.45 (7.61) | 68.93 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 4 | 1 | 5
  Race/Ethnicity: White/Non-Hispanic | 14 | 14 | 28
  Race/Ethnicity: White/Hispanic | 2 | 3 | 5
  Race/Ethnicity: Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Geriatric Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The GAS is a 30 item measure of anxiety symptom severity. The total score is based on a sum of the first 25 items. The remaining 5 items are anxiety content items and are not included in the total score. Total scores range from 0 to 75. Higher scores indicate worse anxiety symptom severity. The measure is a self-report assessment completed at baseline, 4 weeks and 8 weeks.
  units on a scale | 20.85 (8.38) | 22.90 (10.98) | 21.88 (9.70)
Somatic Symptom Scale 8-item [Mean (Standard Deviation); unit: units on a scale] — The Somatic Symptom Scale is an 8-item self-report completed by participant at baseline and 8 weeks. The total score is a sum of the scores for the 8 items on the measure. Measure ranges in total scores from 0 to 32. Higher scores indicate worse somatic symptom severity. Symptoms include stomach/bowel problems, back pain, headaches, etc.
  units on a scale | 9.50 (4.74) | 8.80 (5.63) | 9.15 (5.15)
Patients Health Questionnaire 9-item [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 is a 9 item measure of depressive symptoms. Scores range from 0 to 27. The total score is a sum of the 9 item responses. Higher scores indicate worse depressive symptoms. This measure is a self-report assessment completed at baseline at 8 weeks.
  units on a scale | 8.40 (5.55) | 6.80 (5.48) | 7.60 (5.50)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Symptoms
Description: The Geriatric Anxiety Scale (GAS) is a 30-item measure of somatic, cognitive, and affective symptoms of anxiety. The first 25 items of the measure are used to compute the total score; the last 5 items provide information about the content of worries or fears. Total scores range from 0 to 75 with higher scores indicating worse anxiety. Participants provide severity ratings for items using on a four-point Likert-type scale.
Time Frame: Change from baseline to 8 weeks
Population: A linear mixed effects model using maximum likelihood modeling was employed to analyze these data using intent-to-treat principles.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BREATHE | Wait List
Number analyzed (Participants) | 20 | 20
score on a scale | 17.95 (2.34) | 26.2 (2.14)

2. Primary Outcome: Change in Activity Engagement
Description: The Activity Card Sort contains 80 photographs that depict the performance of instrumental activities, low-physical-demand leisure activities, high-physical-demand leisure activities, and social activities. This measure will be used to assess engagement in activities. The score reported is the lifestyle-adjusted function score. It represents the percentage of activities ever completed that are perceived to be easy. Higher scores indicate greater ease of activity completion/engagement.
Time Frame: Change from baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BREATHE | Wait List
Number analyzed (Participants) | 20 | 19
units on a scale
  Baseline | 49.97 (3.04) | 50.15 (2.83)
  8 weeks | 54.97 (3.57) | 48.23 (3.51)

3. Secondary Outcome: Change in Depressive Symptoms
Description: The Patient Health Questionnaire 9-item (PHQ-9) is a 9-item depression assessment rated on a four-point Likert-type scale with scores ranging from 0 to 27. It includes one item that inquires about suicide ideation. Higher scores indicate more severe depressive symptoms. Validity and reliability have been established with primary care patients.
Time Frame: Change from baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BREATHE | Wait List
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 8.40 (1.24) | 6.80 (1.23)
  8 weeks | 5.71 (1.58) | 8.6 (1.19)

4. Secondary Outcome: Change in Somatic Symptoms
Description: Somatic Symptom Scale (SSS-8). The SSS-8 is an 8-item somatic symptom assessment rated on a five-point Likert-type scale with scores ranging from 0 to 32. The SSS-8 is administered to characterize participants' somatic symptoms. Higher symptoms indicate worse somatic symptom severity.
Time Frame: Change from baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | BREATHE | Wait List
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 9.50 (1.06) | 8.80 (1.26)
  8 weeks | 6.64 (1.07) | 10.30 (1.28)

5. Other Pre Specified Outcome: Change in Heart Rate
Description: Heart rate will be measured at baseline and at 8 weeks after enrollment. This is an exploratory measure.
Time Frame: Change from baseline to 8 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Blood Pressure
Description: Blood pressure will be measured at baseline and at 8 weeks after enrollment. This is an exploratory measure.
Time Frame: Change from baseline to 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: We used the clinicaltrials.gov definition for adverse events reporting. Adverse events were reported via non-systematic assessment. Study assessors and PI were trained to detect any adverse events.
Arm/Group | BREATHE | Wait List
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT02429778/Prot_SAP_000.pdf